CLINICAL TRIAL: NCT04427605
Title: Efficacy and Safety of Continuous Infusion of Ketamine in Pediatric Intensive Care Unit (KISS Study)
Acronym: KISS
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera di Padova (Other)
Responsible Party: Principal Investigator, angela amigoni, Principal Investigator, Azienda Ospedaliera di Padova
Other Study IDs: AOP1795; CESC (Other: Local Ethic Committee for clinical trials)
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Analgesia; Ketamine Toxicity; Bronchospasm; Sedation Complication
Keywords: pediatric intensive care unit; ketamine; sedation
MeSH Terms: conditions — Agnosia; Bronchial Spasm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ketamine group: ketamine intravenous infusion in pediatric patients refractory to conventional analgesic-sedative strategy lasted more than 12 hours (dose range 10-50 mcg/Kg/min)

SUMMARY:
This study, prospectively evaluate the efficacy and safety of ketamine administered in continuous infusion lasted more than 12 hours in children admitted to Pediatric Intensive Care Unit of Padova. This drug may be used as adopted as adopted as adjuvant to analgesia and sedation or as adjuvant to bronchospasm therapy. The investigators evaluated efficacy considering the sparing of other analgesics and sedatives and the level of sedation after ketamine infusion for the first use and the sparing of other bronchospasm drugs sedative dosage for the second use. To evaluate safety the investigators considered the presence of adverse effects and onset of withdrawal and delirium syndrome. The study will included al least 55 pediatric patients < 18 years and mechanically ventilated.

DETAILED DESCRIPTION:
Ketamine is an N-Methyl-d-aspartate-receptor-antagonist commonly used over the last decades as an anesthetic and analgesic agent for procedural sedation. The use of ketamine as a prolonged infusion was first described in 1990 and a prolonged infusion of ketamine has been described as a successful strategy for analgesia and sedation in patients with hemodynamic instability, in patients who were mechanically ventilated and poorly responsive to conventional drugs. An other indication for ketamine infusion is the presence of bronchospasm, due to its action in promoting bronchodilatation. However, existing studies on ketamine for prolonged sedation are mainly retrospective and include small sample size, suggesting that this topic needs to be further investigated. The aim of this observational single center study is to describe the use of ketamine used as adjuvant to conventional analgesic and sedative strategy (opioid and benzodiazepine in continuous infusion) as prolonged infusion (i.e. ≥ 12 hr) in pediatric patients. The investigators will evaluate ketamine indications, dosages, infusion duration, adoption of boluses, modality of weaning. Concomitant analgesic and sedative management and monitoring of level of sedation (using a validated scale) are considered measures of efficacy. Sparing of other bronchospasm drugs sedative dosage are considered measures of efficacy if ketamine is used in patients with obstructive respiratory diseases. Presence of adverse effects (including withdrawal syndrome symptoms and delirium) during infusione or 48 hours after weaning are considered measures of safety. Data were collected using a standardized data sheet. The study lasted 18 months to reach a numerosity of 55 patients. All the requested institutional approvals were collected before starting the data collection.

ELIGIBILITY:
Inclusion Criteria:

* pediatric intensive care unit admission
* mechanical ventilation
* ketamine infusion > 12 hours

Exclusion Criteria:

* parents refusal to participate

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Study population is composed by paediatric patients admitted in PICU treated with ketamine (lasted more than 12 hours) during mechanical ventilation in the studied period.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
level of sedation measured with Comfort Behavior Scale (CBS) | 12 hours
  CBS score decreased > 2 points after ketamine administration

SECONDARY OUTCOMES:
incidence adverse effects,delirium and withdrawal syndrome, assessed by physician (also using Cornell Assessment scale of Pediatric Delirium and Withdrawal Assessment tool 1) | evaluation during all the duration of ketamine infusion till to 48 hours after the end of it
  incidence of adverse effects and number of patients withf delirium (Cornell Assessment scale of Pediatric Delirium) and withdrawal syndrome (Withdrawal Assessment tool 1)
bronchospasm severity | 12 hours
  change of bronchodilator after ketamine infusion

OTHER OUTCOMES:
presence of hypotension | 12 hours
  change of inotropic therapy after ketamine infusion

CONTACTS AND LOCATIONS:
Overall Officials: angela amigoni, MD, Principal Investigator — Azienda Ospedaliera di Padova; andrea pettenazzo, MD, Study Director — Azienda Ospedaliera di Padova
Locations (1):
- Azienda Ospedale Università Padova, Padua, PD, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Heiberger AL, Ngorsuraches S, Olgun G, Luze L, Leimbach C, Madison H, Lakhani SA. Safety and Utility of Continuous Ketamine Infusion for Sedation in Mechanically Ventilated Pediatric Patients. J Pediatr Pharmacol Ther. 2018 Nov-Dec;23(6):447-454. doi: 10.5863/1551-6776-23.6.447. PMID 30697129
- [Background] Zanos P, Moaddel R, Morris PJ, Riggs LM, Highland JN, Georgiou P, Pereira EFR, Albuquerque EX, Thomas CJ, Zarate CA Jr, Gould TD. Ketamine and Ketamine Metabolite Pharmacology: Insights into Therapeutic Mechanisms. Pharmacol Rev. 2018 Jul;70(3):621-660. doi: 10.1124/pr.117.015198. PMID 29945898
- [Background] Miller AC, Jamin CT, Elamin EM. Continuous intravenous infusion of ketamine for maintenance sedation. Minerva Anestesiol. 2011 Aug;77(8):812-20. PMID 21730929
- [Background] Golding CL, Miller JL, Gessouroun MR, Johnson PN. Ketamine Continuous Infusions in Critically Ill Infants and Children. Ann Pharmacother. 2016 Mar;50(3):234-41. doi: 10.1177/1060028015626932. Epub 2016 Jan 18. PMID 26783355
- [Background] Neunhoeffer F, Hanser A, Esslinger M, Icheva V, Kumpf M, Gerbig I, Hofbeck M, Michel J. Ketamine Infusion as a Counter Measure for Opioid Tolerance in Mechanically Ventilated Children: A Pilot Study. Paediatr Drugs. 2017 Jun;19(3):259-265. doi: 10.1007/s40272-017-0218-4. PMID 28299720
- [Background] Allen JY, Macias CG. The efficacy of ketamine in pediatric emergency department patients who present with acute severe asthma. Ann Emerg Med. 2005 Jul;46(1):43-50. doi: 10.1016/j.annemergmed.2005.02.024. PMID 15988425
- [Background] Petrillo TM, Fortenberry JD, Linzer JF, Simon HK. Emergency department use of ketamine in pediatric status asthmaticus. J Asthma. 2001 Dec;38(8):657-64. doi: 10.1081/jas-100107543. PMID 11758894